CLINICAL TRIAL: NCT03646058
Title: Add-on Buprenorphine at Analgesic Doses for the Treatment of Severe Suicidal Ideas During a Major Depressive Episode
Acronym: BUPRIS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC-N/2017/FJ-01
Record Dates: First submitted 2018-08-16; First posted 2018-08-24 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Suicidal Ideation; Major Depressive Episode
Keywords: Treatment; Suicidal ideas; Depression; Buprenorphine; Opioid agonist; Mental pain
MeSH Terms: conditions — Suicidal Ideation; Depression | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): 2 placebo pills sublingual during 28 days
  Interventions: Drug: Placebo
- 0.4mg buprenorphine (Experimental): 1 pill of 0.4 mg buprenorphine + 1 placebo pill per day for 21 days, then 2 placebo pills per day for 1 week, all sublingual.
  Interventions: Drug: Buprenorphine
- 0.8mg buprenorphine (Experimental): 1 pill of 0.4 mg buprenorphine + 1 placebo pill per day for 3 days, then 2 pills of 0.4mg buprenorphine per day for 18 days, then 1 pill of 0.4 mg + 1 placebo pill per day for 3 days, then 2 placebo pills per day for 4 days, all sublingual.
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — Buprenorphine, 0.4mg pills, sublingual
  Other Names: Temgesic
  Arms: 0.4mg buprenorphine; 0.8mg buprenorphine
Drug: Placebo — Placebo pills, sublingual, specifically made to mimick buprenorphine pills
  Arms: Placebo

SUMMARY:
This study aims at investigating if adjunctive buprenorphine at low dose to treatment as usual is effective in reducing severe suicidal ideas in major depressive episode, and at determining the most effective dose.

DETAILED DESCRIPTION:
Participants will be randomized to two doses of buprenorphine (0.4mg and 0.8mg) or placebo. The duration of treatment will be 21 days with 7 days withdrawal period. Two follow-up phone calls at 3 and 6 months will investigate occurence of suicidal behavior.

The main outcome will be changes in suicidal ideas levels during the first week.

Secondary outcomes will be changes in suicidal ideas during the following 21 days, changes in depression and psychological pain levels over the first 28 days, dropout rates, reasons and occurence of side effects over the first 28 days, withdrawal symptoms dung the withdrawal period, changes in neuropsychological and neuroimaging measures between Day 0 and Day 28.

Blood and stool samples will be collected at 4 time points and stored in a biobank for future analyses.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been correctly informed.
* The patient must have given his/her informed and signed the consent form.
* The patient must be insured or beneficiary of a health insurance plan.
* The patient is at least 18 years old and 65 years old at the most.
* The patient is hospitalized or followed in consultation.
* The patient has a current major depressive episode without psychotic features according to the criteria of the "Diagnostic and Statistical Manual of Mental Disorders"
* The patient has a score > 20 of the "Montgomery-Asberg Depression Rating Scale".
* The patient has a current Scale for Suicidal Ideation (SSI) score > 8.

Exclusion Criteria:

* The patient is participating in another interventional trial;
* The patient is in an exclusion period determined by a previous study;
* The patient is under judicial protection, or is an adult under guardianship;
* The patient is under compulsory admission;
* The patient refuses to sign the consent;
* it is impossible to correctly inform the patient.
* The patient is pregnant or breastfeeding.
* The patient suffers from schizophrenia;
* The patient suffered from moderate to severe alcohol use disorder or substance use disorder (except tobacco and caffeine) over the last 12 months according to DSM-5 criteria ;
* The patient currently suffers from severe and/or unstable medical condition (including severe respiratory or hepatic insufficiency) or a painful medical condition;
* The patient has a current known sleep apnea.
* The patient currently takes analgesic treatment (including Nonsteroidal anti-inflammatory drug and paracetamol);
* The patient currently takes central nervous depressant drugs at sedative doses (based on the investigator's assessment), including benzodiazepines, antihistamines, and sedative antipsychotics;
* The patient currently takes major CYP3A4 Inhibitors and inducers;
* The patient currently takes has received Electroconvulsivotherapy over the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Beck Scale for Suicidal Ideation (SSI) scores from Day 0 to 7 | 7 days
  Clinician-based questionnaire measuring level of suicidal ideas over the last 7 days; 21 items scored 0 to 2; total score ranges from 0 to 38 (last 2 items not counted), higher scores mean more intense suicidal ideas.

SECONDARY OUTCOMES:
Changes in Beck Scale for Suicidal Ideation (SSI) scores | Day 8 to day 28
  Clinician-based questionnaire measuring level of suicidal ideas over the last 7 days; 21 items scored 0 to 2; total score ranges from 0 to 38 (last 2 items not counted); higher scores mean more intense suicidal ideas.
Changes in Beck Depression Inventory II (BDI-II) scores from Day 0 to 28 | 28 days
  Self questionnaire measuring depression level over the last 7 days; 13 items scored 0 to 3, with the total score ranging from 0 to 39; higher scores mean higher level of depression.
Changes in Montgomery-Asberg Depression Rating Scale (MADRS) from Day 0 to 28 | 28 days
  Clinician-based questionnaire measuring the level of depression of the last 7 days; 10 items score 0 to 6, with the total scores ranging fron 0 to 60; Higher scores mean higher level of depression.
Changes in Physical and Psychological Pain - Visual Analog Scale (PPP-VAS) scores from Day 0 to 28 | 28 days
  Visual Analog Scale measuring physical then psychological pain over 3 periods each (current, worst over the last 7 days, mean over the last 7 days); 6 dimensions in total; each dimension is scored from 0 (no pain) to 10 (maximal pain).
Reasons for discontinuing treatment over the first 28 days | 28 days
  Patient's self-report; measurement will be the overall (over 28 days) incidence for each event reported.
Side effects over the first 28 days | 28 days
  Patient's self-report; measurement will be the overall (over 28 days) incidence for each event reported.
Withdrawal symptoms | Day 22 to day 28
  Patient's self-report; measurement will be the incidence of any withdrawal symptom during the withdrawal phase.
Occurence of a suicide attempt during the whole study | 180 days
  Interview based; measurement will be the incidence of any suicide attempt between Day 0 and 28, between Day 29 and 90, and between Day 90 and 180.
Changes in Iowa Gambling Task (IGT) scores between Day 0 and 28 | 28 days
  Computerized test measuring decision-making; scores are the difference between advantageous and disadvantageous choices; scores range from -100 to + 100, higher scores means better performance
Changes in modified Stroop test scores between Day 0 and 28 | 28 days
  Classical Stroop test modified with suicide-related words to measure specific attention bias; scores are the number of errors and total reaction time; higher scores mean worse performance
Changes in verbal fluency test scores between Day 0 and 28 | 28 days
  Classical test measuring verbal fluency skills for semantic and phonological categories; Patients are instructed to give as many words as possible for a given category then for words starting with a given letter, within a 1 minute time frame; Scores are the number of correct words; higher scores mean higher performance
Changes in N-Back test scores between Day 0 and 28 | 28 days
  Classical test of working memory using letters; scores are the number of words correctly identified for each level of recall (0 to 2 back); higher scores mean better performance; also, the number of omission and commission errors.
Changes in Go/No-Go test between Day 0 and 28 | 28 days
  Classical test of cognitive inhibition, letter version; scores are the number of omission and commission errors (higher scores mean worse performance) and reaction times (higher scores mean better performance)
Changes in Trail Making Test (TMT) scores between Day 0 and 28 | 28 days
  Classical test of planning abilities; scores are the difference between the time to complete parts B and A of the test; Higher scores mean worse performance.
Changes in Implicit Association Test (IAT) scores between Day 0 and 28 | 28 days
  IAT version adapted for suicide/death; scores are the measure of reaction times in the association between suicide/death words and me/myself words; lower scores mean higher association.
Changes in Magnetic Resonance Imaging (MRI) T1 measures between Day 0 and 28 | 28 days
  Brain structural MRI-T1 sequence measured at Day 0 and Day 28 (5 minutes)
Changes in Magnetic Resonance Imaging (MRI) T2 measures between Day 0 and 28 | 28 days
  Brain structural MRI-T2 sequence measured at Day 0 and Day 28 (5 minutes)
Changes in Magnetic Resonance Imaging (MRI) Diffusion Tensor Imaging (DTI) measures between Day 0 and 28 | 28 days
  Brain Diffusion Tensor Imaging (DTI) sequence measured at Day 0 and Day 28 (20 minutes)
Changes in Magnetic Resonance Imaging (MRI) Resting State (RS) measures between Day 0 and 28 | 28 days
  Brain functional Resting State (RS) sequence measured at Day 0 and Day 28 (15 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Jollant, MD, Principal Investigator — Hôpital Sainte-Anne
Locations (9):
- France (9):
  - Ch Perrens, Bordeaux, France
  - CHU Bicêtre, Le Kremlin-Bicêtre
  - Hospices Civils de Lyon, Lyon
  - CAPPA Jacques PREVERT, Nantes
  - CHU Nîmes, Nîmes
  - CH Sainte-Anne, Paris
  - CH Henri Laborit, Poitiers
  - Chu Toulouse Hopital Purpan, Toulouse
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No